CLINICAL TRIAL: NCT00055965
Title: A Pragmatic, Randomised Study To Compare The Hospitalisation Rates Of Two Platinum-Based Outpatient Regimens (Gemcitabine/Cisplatin vs. Gemcitabine/Carboplatin) In Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Hospitalization Rates of Patients With Non-Small Cell Lung Cancer Treated With Gemcitabine and Either Cisplatin or Carboplatin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000271903; CHNT-GEM-HOSP; EU-20245
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-01

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Cisplatin; Gemcitabine

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known if one regimen will require patients to spend more time in the hospital than the other regimen for treatment of chemotherapy-related side effects.

PURPOSE: Randomized phase III trial to compare the hospitalization rates of patients who are receiving gemcitabine combined with cisplatin with that of patients receiving gemcitabine combined with carboplatin for unresectable stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the rates of overnight hospitalization due to toxicity (e.g., blood transfusion, antibiotic use, and to obtain relief of treatment-related symptoms) of patients with non-small cell lung cancer treated with gemcitabine and cisplatin vs gemcitabine and carboplatin.
* Compare the need for hospitalization for chemotherapy administration in patients treated with these regimens.
* Compare the tumor response rate of patients treated with these regimens.
* Compare the overall survival of patients treated with these regimens.
* Compare the relief of tumor-related symptoms in patients treated with these regimens.
* Compare the effect on Karnofsky performance status in patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to stage (IIIA vs IIIB [dry] vs IIIB [wet] or IV) and performance status (50-60% vs 70-100%). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes and cisplatin IV over 1-2 hours on days 1 and 8.
* Arm II: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and carboplatin IV over 30-60 minutes on day 1.

In both arms, treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 6 months and then every 3-4 months thereafter.

PROJECTED ACCRUAL: A total of 400 patients (200 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed inoperable non-small cell lung cancer

  * Stage IIIA, IIIB, or IV
  * Not eligible for curative radiotherapy or surgery
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 50-100%

Life expectancy

* At least 12 weeks

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 3 times ULN (5 times ULN if liver metastases present)

Renal

* Creatinine no greater than ULN OR
* Creatinine clearance at least 60 mL/min

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after study completion
* No active infection
* No serious systemic disorder that would preclude study participation
* No grade 2 or greater peripheral neuropathy
* No significant neurological problems (e.g., seizures or psychiatric disorders)
* No other active malignancy within the past 5 years except carcinoma in situ of the cervix or adequately treated non-melanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior cytotoxic chemotherapy
* No other concurrent chemotherapy during or for 7 days after study therapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy
* No concurrent radiotherapy during or for 7 days after study therapy

Surgery

* See Disease Characteristics

Other

* At least 12 weeks since prior investigational agents
* No other concurrent antitumor therapy
* No concurrent experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2002-11; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Rate of hospitalization due to toxicity

SECONDARY OUTCOMES:
Need for hospitalization for chemotherapy administration
Tumor response rate
Overall survival
Relief of tumor-related symptoms
Effect on Karnofsky performance status
Toxicity as measured by NCIC CTC v2.0

CONTACTS AND LOCATIONS:
Overall Officials: Nick Thatcher, PhD, FRCP, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- Christie Hospital NHS Trust, Manchester, England, United Kingdom